CLINICAL TRIAL: NCT00476983
Title: Pharmacokinetic and Efficacy of Saquinavir Mesylate Film Coated Tablet / Ritonavir 1500/100 Plus Tenofovir/Emtricitabine 300/200 mg Once Daily in HIV Pretreated Patients
Brief Title: Pharmacokinetic and Efficacy of SQV/r 1500/100 Plus Tenofovir/Emtricitabine 300/200 mg
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No funding
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 041
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Saquinavir/Ritonavir BID or Lopinavir/Ritonavir BID
Keywords: saquinavir/ritonavir 1500/100 mg once daily
MeSH Terms: interventions — Saquinavir; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): SQV/r 1500/100 mg OD + Truvada OD
  Interventions: Drug: saquinavir/ritonavir plus truvada

INTERVENTIONS:
Drug: saquinavir/ritonavir plus truvada — SQV/r 1500/100 mg OD + Truvada OD for 2 years

SUMMARY:
Pharmacokinetic and long term efficacy of TDF SQV film coated tablet 1500/100mg once daily plus TDF/FTC300/200mg once daily.

DETAILED DESCRIPTION:
This study will be performed in patients who were previously treated with SQV /r 1000/100mg twice daily or Lopinavir/r plus TDF/FTC once daily as part of the Gemini study. After 48 weeks of the study, the patients will be treated with SQV film coated tablet 1500/100mg once daily plus TDF/FTC300/200mg once daily with good CD4 and VL outcomes. In this study, we would like to evaluate the once-daily dosing of SQV using SQV- SQV film coated tablet 1500/ritonavir 100mg in combination with TDF/FTC300/200mg once daily. We believe that the PK parameters of SQV given at 1500mg daily will be equivalent to the 1000mg twice daily dosing when combined with RTV and TDF/FTC300/200mg OD, and that the once daily regimen will have better safety, tolerability profile than the twice daily regimen while maintaining good CD4 and VL outcome

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent
2. All adults HIV patients previously included in the Gemini study and are currently enrolled in HIV-NAT 006 and treated with SQV /r 1500/100 mg OD plus tenofovir/emtricitabine (TDF/FTC) 300/200 mg once daily

Exclusion Criteria:

1. Inability to understand the nature and extent of the study and the procedures required.
2. ALT/ AST more than 5x upper limit
3. Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion.
4. Use of concomitant medication that may interfere with the pharmacokinetics of saquinavir, ritonavir, tenofovir or emtricitabine
5. History of sensitivity/idiosyncrasy to the drug or chemically related compounds which may be employed in the study.
6. Active drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of saquinavir mesylate film-coated tablet 1500 mg once daily dosing when used in combination with ritonavir 100 mg, and tenofovir/emtricitabine (TDF/FTC) 300/200 mg once daily | 96 weeks

SECONDARY OUTCOMES:
safety, tolerability and efficacy of SQV /r 1500/100 once daily when use with TDF/FTC | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT)

REFERENCES:
- See also: The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org